CLINICAL TRIAL: NCT02573129
Title: Effects of Incorporating Red Meat Into a Mediterranean-style Dietary Pattern on Cardiometabolic and Emotional Well-being
Brief Title: The Lean Meats Mediterranean Diet Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Pork Board (Other); National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PurdueU
Record Dates: First submitted 2015-05-28; First posted 2015-10-09 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular Diseases; Dietary Modification
Keywords: cardiovascular disease risk; Mediterranean diet; red meat
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red Meat Restricted (Experimental): Following a 2-wk baseline testing period to assess cardiometabolic and emotional well-being and habitual diet, subjects will consume a Mediterranean-style, weight-maintenance diet that is restricted in lean, minimally processed red meat for 5 weeks.
  Interventions: Other: Red Meat Restricted; Other: Red Meat Rich
- Red Meat Rich (Experimental): Following a 4-wk wash out period and a 2-wk baseline testing period to assess cardiometabolic and emotional well-being and habitual diet, subjects will consume a Mediterranean-style, weight-maintenance diet that is rich in lean, minimally processed red meat for 5 weeks.
  Interventions: Other: Red Meat Restricted; Other: Red Meat Rich

INTERVENTIONS:
Other: Red Meat Restricted — restrict intake of red meat while a Mediterranean diet
  Other Names: S44 Mediterranean Diet
Other: Red Meat Rich — Mediterranean diet rich in red meat
  Other Names: S44 Mediterranean Diet

SUMMARY:
The purpose of the proposed research study is to assess the effects of including greater amounts of minimally processed red meat (lean pork and beef) into a Mediterranean Diet on cardiometabolic and emotional well-being.

DETAILED DESCRIPTION:
All subjects will complete an 18-wk randomized crossover study. Following a 2-wk baseline testing period to assess cardiometabolic and emotional well-being and habitual diet, subjects will consume a Mediterranean-style, weight-maintenance diet that is either restricted or rich in lean, minimally processed red meat for 5 weeks. Following a 4-wk washout period and second 2-wk baseline testing, subjects will consume the Mediterranean Diet with the alternate predominant animal protein sources for 5 weeks. Cardiometabolic and emotional well-being will be assessed during baseline and post periods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 30-69 years old
* BMI 25-37 kg/m2
* Total cholesterol <240 mg/dL
* Low-density lipoprotein <160 mg/dL
* Triglycerides <400 mg/dL
* Fasting glucose <110 mg/dL
* Systolic blood pressure <160 mmHg
* Diastolic blood pressure <100 mmHg
* Body weight <300 lb
* Weight stable for 3 months prior (±10 lb)
* Stable physical activity regimen 3 months prior ≤3 h/wk of moderate or high intensity exercise resistance or aerobic training
* Medication use stable for 6 months prior.

Exclusion Criteria:

* Diabetic
* Smoker

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
blood pressure | 5 weeks
  clinical and 24-hr monitoring
lipid profile | 5 weeks
  cholesterol panel

SECONDARY OUTCOMES:
sleep quality | 5 weeks
  sleep assessed by using actigraphy / actiwatch
sleep assessment | 5 wks
  Sleep assessed by questionnaires using the Pittsburgh Sleep Quality Index
assessment of sleep | 5 weeks
  Sleep assessed by questionnaires using the SF-36v2® Health Survey
emotional well-being | 5 weeks
  quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wayen W Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University - Stone Hall 700 W State St, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Hill EB, Reisdorph RM, Rasolofomanana-Rajery S, Michel C, Khajeh-Sharafabadi M, Doenges KA, Weaver N, Quinn K, Sutliff AK, Tang M, Borengasser SJ, Frank DN, O'Connor LE, Campbell WW, Krebs NF, Hendricks AE, Reisdorph NA. Salmon Food-Specific Compounds and Their Metabolites Increase in Human Plasma and Are Associated with Cardiometabolic Health Indicators Following a Mediterranean-Style Diet Intervention. J Nutr. 2024 Jan;154(1):26-40. doi: 10.1016/j.tjnut.2023.10.024. Epub 2023 Oct 31. PMID 37918675
- [Derived] O'Connor LE, Biberstine SL, Paddon-Jones D, Schwichtenberg AJ, Campbell WW. Adopting a Mediterranean-Style Eating Pattern with Different Amounts of Lean Unprocessed Red Meat Does Not Influence Short-Term Subjective Personal Well-Being in Adults with Overweight or Obesity. J Nutr. 2018 Dec 1;148(12):1917-1923. doi: 10.1093/jn/nxy235. PMID 30517731
- [Derived] O'Connor LE, Paddon-Jones D, Wright AJ, Campbell WW. A Mediterranean-style eating pattern with lean, unprocessed red meat has cardiometabolic benefits for adults who are overweight or obese in a randomized, crossover, controlled feeding trial. Am J Clin Nutr. 2018 Jul 1;108(1):33-40. doi: 10.1093/ajcn/nqy075. PMID 29901710